CLINICAL TRIAL: NCT02015663
Title: A 24-week, Open-label, Parallel-group, Interventional Phase IV Study Comparing Tobramycin Inhalation Powder (TIP) Administered Once Daily Continuously Versus TIP Administered BID in 28 Day on / 28 Day Off Cycles for the Treatment of Pulmonary Pseudomonas Aeruginosa in Patients With Cystic Fibrosis
Brief Title: Tobramycin Inhalation Powder (TIP) Administered Once Daily Continuously Versus TIP Administered BID in 28 Day on / 28 Day Off Cycles
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CTBM100CUS03
Record Dates: First submitted 2013-12-13; First posted 2013-12-19 (Estimated); Results first posted 2017-03-29 (Actual); Last update posted 2017-03-29 (Actual); Status verified 2017-02

CONDITIONS: Cystic Fibrosis
Keywords: Cystic Fibrosis; CF
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Experimental): Tobramycin Inhalation Powder (112 mg) once daily during 168 days
  Interventions: Drug: Tobramycin Inhalation Powder
- Arm 2 (Active Comparator): Tobramycin Inhalation Powder (112 mg) twice daily on days 1-28, days 57-84 and days 113-140
  Interventions: Drug: Tobramycin Inhalation Powder

INTERVENTIONS:
Drug: Tobramycin Inhalation Powder — Tobramycin Inhalation Powder 112 mg (four 28-mg capsules) taken via inhaler once or twice a day, depending on study arm

SUMMARY:
To provide efficacy and safety data comparing two dosing schedules of Tobramycin Inhalation Powder (TIP) for the treatment of pulmonary Pseudomonas aeruginosa in patients with cystic fibrosis.

ELIGIBILITY:
Inclusion Criteria:

1. Provide written informed consent, HIPPA (Health Insurance Portability and Accountability Act) authorization (where applicable), and assent (as appropriate) prior to the performance of any study-related procedure.
2. Confirmed diagnosis of CF
3. FEV1 at screening (Visit 1) ≥25% and ≤ 80% of normal predicted values for age, sex, and height
4. P. aeruginosa must be present within 6 months prior to screening and at screening
5. Able to comply with all protocol requirements
6. Clinically stable in the opinion of the investigator

Exclusion Criteria:

1. History of Burkholderia cenocepacia (Bcc) complex within 2 years prior to screening and/or Bcc complex at screening
2. Hemoptysis more than 60 cc at any time within 30 days prior to study drug administration
3. History of hearing loss or chronic tinnitus deemed clinically significant by the investigator
4. Serum creatinine 2 mg/dL or greater, BUN 40 mg/dL or greater, or an abnormal urinalysis defined as 2+ or greater proteinuria at screening
5. Known local or systemic hypersensitivity to aminoglycosides or inhaled antibiotics
6. Patients who are unable to discontinue previously received inhaled antibiotic regimen(s) (inhaled antibiotics are not allowed other than study drug)
7. Use of inhaled aminoglycosides within 28 days prior to study drug administration (Visit 2)
8. Use of systemic anti-pseudomonal antibiotics within 28 days prior to study drug administration
9. Use of loop diuretics within 7 days prior to study drug administration
10. Administration of any investigational drug within 30 days prior to enrollment or 5 half-lives, whichever is longer
11. Signs and symptoms of acute pulmonary disease, e.g , pneumonia, pneumothorax
12. Hospitalization during the baseline visit
13. History of malignancy
14. Patients with clinically significant laboratory abnormalities (not associated with the study indication) at screening
15. Patients with other clinically significant conditions (not associated with the study indication) which might interfere with the assessment of this study
16. Patients or caregivers with a history of noncompliance to medical regimens and patients or caregivers who are considered potentially unreliable
17. Pregnant or nursing (lactating) women
18. Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, including women whose career, lifestyle, or sexual orientation precludes intercourse with a male partner and women whose partners have been sterilized by vasectomy or other means, UNLESS they are using two birth control methods.

Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2014-01; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (21):
- United States (21):
  - Novartis Investigative Site, Mobile, Alabama
  - Novartis Investigative Site, Los Angeles, California
  - Novartis Investigative Site, Sacramento, California
  - Novartis Investigative Site, Ventura, California
  - Novartis Investigative Site, Altamonte Springs, Florida
  - Novartis Investigative Site, Jacksonville, Florida
  - Novartis Investigative Site, Miami, Florida
  - Novartis Investigative Site, Orlando, Florida
  - Novartis Investigative Site, Pensacola, Florida
  - Novartis Investigative Site, Glenview, Illinois
  - Novartis Investigative Site, Indianapolis, Indiana
  - Novartis Investigative Site, Iowa City, Iowa
  - Novartis Investigative Site, St Louis, Missouri
  - Novartis Investigative Site, New Hyde Park, New York
  - Novartis Investigative Site, New York, New York
  - Novartis Investigative Site, Akron, Ohio
  - Novartis Investigative Site, Oklahoma City, Oklahoma
  - Novartis Investigative Site, Portland, Oregon
  - Novartis Investigative Site, Hershey, Pennsylvania
  - Novartis Investigative Site, Austin, Texas
  - Novartis Investigative Site, Salt Lake City, Utah

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study intended to randomize 200 patients in 18 months; however, after 9 months, only 25 patients were randomized, with a screen fail rate of 50%. Due to premature termination, summaries and analyses planned in the protocol were eliminated in the statistical analysis plan prior to database lock. No inferential analysis will be provided.
Groups:
- Tobramycin Inhalation Powder Once Daily: Tobramycin Inhalation Powder (112 mg) once daily during 168 days
- Tobramycin Inhalation Powder Twice Daily: Tobramycin Inhalation Powder (112 mg) twice daily on days 1-28, days 57-84 and days 113-140
Period: Overall Study
Arm/Group | Tobramycin Inhalation Powder Once Daily | Tobramycin Inhalation Powder Twice Daily
Started | 16 | 16
Completed | 1 | 4
Not Completed | 15 | 12
Not completed — unsatisfactory therapeutic effect | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Protocol Violation | 0 | 1
Not completed — Adverse Event | 3 | 0
Not completed — Administrative problems | 10 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tobramycin Inhalation Powder Once Daily | Tobramycin Inhalation Powder Twice Daily | Total
Number analyzed (Participants) | 16 | 16 | 32
Age, Continuous [Mean (Standard Deviation); unit: year] | 34.9 (14.31) | 26.5 (11.09) | 30.7 (13.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 8 | 14
  Male | 10 | 8 | 18

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Forced Expiratory Volume in 1 Second ( FEV1) Percent Predicted
Description: The Forced Expiratory Volume in 1 second (FEV1) percent predicted expresses FEV1 as a percentage of the "predicted values" for participants of similar characteristics (height, age, sex, and sometimes race and weight). A positive change from baseline in FEV1 percent predicted indicates improvement in lung function.
Time Frame: Baseline and Day 168
Population: The study intended to randomize 200 patients within 18 months; however, after 9 months, only 32 patients were successfully randomized, with a screen fail rate of 50%. Study was terminated with only safety data analyzed. No data collected met the pre-specified powering of 200 patients needed for analysis (only 32 patients randomized)
Arm/Group | Tobramycin Inhalation Powder Once Daily | Tobramycin Inhalation Powder Twice Daily
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Percent Change From Baseline in Forced Expiratory Volume in 1 Second (FEV1) Percent Predicted
Description: as for outcome 1
Time Frame: Baseline and Day 168
Population: as for outcome 1
Arm/Group | Tobramycin Inhalation Powder Once Daily | Tobramycin Inhalation Powder Twice Daily
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Percent Change From Baseline in Forced Vital Capacity (FVC) Percent Predicted
Description: Forced Vital Capacity (FVC) is the amount of air which can be forcibly exhaled from the lungs after taking the deepest breath possible. FVC will be assessed via spirometry. A positive change from baseline in FVC indicates improvement in lung function.
Time Frame: Baseline and Day 168
Population: as for outcome 1
Arm/Group | Tobramycin Inhalation Powder Once Daily | Tobramycin Inhalation Powder Twice Daily
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Percent Change From Baseline in Forced Expiratory Flow (FEF) 25%-75% Predicted
Description: The Forced Expiratory Flow (FEF) 25%-75% measurement describes the amount of air expelled from the lungs during the middle half (25% - 75%) of the forced vital capacity test and is measured using spirometry. A positive change from baseline in FEF indicates improvement in lung function. The predicted percent will be assessed.
Time Frame: Baseline and day 168
Population: as for outcome 1
Arm/Group | Tobramycin Inhalation Powder Once Daily | Tobramycin Inhalation Powder Twice Daily
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Change From Baseline in Pseudomonas Aeruginosa Sputum Density
Description: Change from baseline in Pseudomonas aeruginosa sputum density will be measured by log10 colony forming units per gram of sputum.
Time Frame: Baseline and day 168
Population: as for outcome 1
Arm/Group | Tobramycin Inhalation Powder Once Daily | Tobramycin Inhalation Powder Twice Daily
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Time to First Hospitalization Due to Respiratory-related Events
Description: Time to the first hospitalization due to respiratory-related events (number of days) per patient.
Time Frame: Day 1 to day 168
Population: as for outcome 1
Arm/Group | Tobramycin Inhalation Powder Once Daily | Tobramycin Inhalation Powder Twice Daily
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Percentage of Patients With Hospitalizations Due to Respiratory-related Events
Description: Percentage of patients with hospitalization due to respiratory-related events
Time Frame: Day 1 to day 168
Population: as for outcome 1
Arm/Group | Tobramycin Inhalation Powder Once Daily | Tobramycin Inhalation Powder Twice Daily
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Length of Hospital Stay Due to Respiratory-related Events
Description: The number of days in length of hospital stay per patient due to respiratory-related events will be measured.
Time Frame: Day 1 to day 168
Population: as for outcome 1
Arm/Group | Tobramycin Inhalation Powder Once Daily | Tobramycin Inhalation Powder Twice Daily
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Time to First Usage of Anti-pseudomonal Antibiotic
Description: Time to first usage of anti-pseudomonal antibiotic per patient will be assessed by number of days
Time Frame: Day 1 to day 168
Population: as for outcome 1
Arm/Group | Tobramycin Inhalation Powder Once Daily | Tobramycin Inhalation Powder Twice Daily
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Percentage of Patients Who Use Anti-pseudomonal Antibiotic
Description: Percentage of patients who use anti-pseudomonal antibiotic will be assessed.
Time Frame: Day 1 to day 168
Population: as for outcome 1
Arm/Group | Tobramycin Inhalation Powder Once Daily | Tobramycin Inhalation Powder Twice Daily
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Duration of Use of Anti-pseudomonal Antibiotic
Description: Number of days of use of anti-pseudomonal antibiotic per patient will be assessed.
Time Frame: Day 1 to day 168
Population: as for outcome 1
Arm/Group | Tobramycin Inhalation Powder Once Daily | Tobramycin Inhalation Powder Twice Daily
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Change From Baseline in Tobramycin Minimal Inhibitory Concentration for Pseudomonas Aeruginosa
Description: Change from baseline in tobramycin minimal inhibitory concentration for Pseudomonas aeruginosa will be measured by laboratory testing.
Time Frame: Baseline and day 168
Population: as for outcome 1
Arm/Group | Tobramycin Inhalation Powder Once Daily | Tobramycin Inhalation Powder Twice Daily
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Tobramycin Inhalation Powder Once Daily | Tobramycin Inhalation Powder Twice Daily | Total Events
Serious Adverse Events (participants affected / at risk) | 3/16 | 1/15 | 4/31
Other Adverse Events (participants affected / at risk) | 13/16 | 12/15 | 25/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tobramycin Inhalation Powder Once Daily (N=16) | Tobramycin Inhalation Powder Twice Daily (N=15) | Total Events (N=31)
Infective pulmonary exacerbation of cystic fibrosis (Infections and infestations) | 2 | 1 | 3
Endometriosis (Reproductive system and breast disorders) | 1 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tobramycin Inhalation Powder Once Daily (N=16) | Tobramycin Inhalation Powder Twice Daily (N=15) | Total Events (N=31)
Palpitations (Cardiac disorders) | 0 | 1 | 1
Hypoacusis (Ear and labyrinth disorders) | 1 | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 2 | 1 | 3
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 2 | 1 | 3
Abdominal pain upper (Gastrointestinal disorders) | 0 | 2 | 2
Constipation (Gastrointestinal disorders) | 1 | 1 | 2
Diarrhoea (Gastrointestinal disorders) | 2 | 1 | 3
Dry mouth (Gastrointestinal disorders) | 0 | 1 | 1
Nausea (Gastrointestinal disorders) | 3 | 0 | 3
Post-tussive vomiting (Gastrointestinal disorders) | 0 | 1 | 1
Vomiting (Gastrointestinal disorders) | 1 | 1 | 2
Asthenia (General disorders) | 1 | 2 | 3
Chest discomfort (General disorders) | 2 | 0 | 2
Chills (General disorders) | 0 | 1 | 1
Fatigue (General disorders) | 1 | 1 | 2
Pain (General disorders) | 0 | 2 | 2
Pyrexia (General disorders) | 1 | 1 | 2
Drug hypersensitivity (Immune system disorders) | 1 | 0 | 1
Infective pulmonary exacerbation of cystic fibrosis (Infections and infestations) | 0 | 4 | 4
Otitis media (Infections and infestations) | 1 | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 0 | 1
Anaemia postoperative (Injury, poisoning and procedural complications) | 1 | 0 | 1
Gastrointestinal disorder postoperative (Injury, poisoning and procedural complications) | 1 | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 1 | 0 | 1
Vaccination complication (Injury, poisoning and procedural complications) | 1 | 0 | 1
Hepatic enzyme increased (Investigations) | 1 | 0 | 1
Liver function test abnormal (Investigations) | 0 | 1 | 1
Oxygen saturation decreased (Investigations) | 0 | 1 | 1
Pulmonary function test decreased (Investigations) | 3 | 1 | 4
Weight decreased (Investigations) | 1 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Benign ovarian tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Aphonia (Nervous system disorders) | 1 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 2 | 2
Dysgeusia (Nervous system disorders) | 0 | 1 | 1
Neuralgia (Nervous system disorders) | 0 | 1 | 1
Anxiety (Psychiatric disorders) | 0 | 2 | 2
Depression (Psychiatric disorders) | 0 | 1 | 1
Cervical dysplasia (Reproductive system and breast disorders) | 1 | 0 | 1
Fallopian tube cyst (Reproductive system and breast disorders) | 1 | 0 | 1
Haemorrhagic ovarian cyst (Reproductive system and breast disorders) | 1 | 0 | 1
Ovarian cyst (Reproductive system and breast disorders) | 1 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 10 | 9 | 19
Dry throat (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 5
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 3
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 4
Pharyngeal oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Prolonged expiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Rhonchi (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 3
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 1

LIMITATIONS AND CAVEATS:
Due to premature termination, summaries and analyses planned in the protocol were eliminated in the statistical analysis plan prior to database lock. No inferential analysis will be provided.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.